CLINICAL TRIAL: NCT06310928
Title: The Effect of Thermal Blanket Applied to the Area After Peripheral Artery Surgery on Circulation, Pain and Mobilization
Brief Title: The Effect of Thermal Blanket After Peripheral Artery Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, SONAY GÖKTAŞ, Prof.Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SBU-201001077-2022
Record Dates: First submitted 2024-02-13; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Peripheral Arterial Disease
Keywords: Thermal Blanket; Effect; Pain; Mobilization; Circulation
MeSH Terms: conditions — Peripheral Arterial Disease; Pain

STUDY DESIGN:
Intervention Model Description: This study is a single center randomized controlled clinical trial.The sample consisted of a total of 60 patients who would undergo interventional peripheral arterial surgery, met the study criteria and agreed to participate in this study. They will be divided into two groups as 30 experimental group and 30 control group by randomization method.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermal Blanket Intervention Group (Experimental): After the informed consent form is signed by the patients, general body warming of the patient will be provided with the hot air blowing system after surgery. In the 30th minute of the active heating method, a thermal blanket will be applied to the treated area (extremity) of the patient. The first 24 hours after the application; Pain will be evaluated every hour for the first 8 hours, every 2 hours for the second 8 hours, every 4 hours for the last 8 hours with the VAS Pain Scale and circulation with the Neurovascular Diagnosis Form. Mobilization of the patient for the first time in the 8th hour and for the second time in the 24th hour will be evaluated with the Patient and Observer Mobility Scale. Pain and neurovascular evaluation will be performed every 12 hours on the second postoperative day. Mobility will be assessed for the third time on the second postoperative day.
  Interventions: Other: Thermal Blanket
- Control Group (No Intervention): After the informed consent form was signed by the patients who agreed to participate in the study before the application and who met the inclusion criteria, respectively;The vital signs of patients admitted to the intensive care unit after surgery will be stabilized.The patient's general warming of the body will be ensured with the hot air blowing system (Forced-air), which is an active heating method.Afterwards, the treated extremity will be wrapped with cotton alban, which is a routine application.Tests will be performed to the participants in the control group at the same time as in the experimental group.

INTERVENTIONS:
Other: Thermal Blanket — Thermal blankets, a passive heating blanket, have a silver surface to prevent heat loss through radiation. Thermal insulation is achieved thanks to the fact that they are covered with a reflective surface to reflect light radiation, i.e. thermal radiation. It is a cost-effective, easy-to-clean, flexible material that takes the desired shape. Thermal blankets generate heat by providing thermal insulation with infrared radiation and can provide thermal vasodilation or thermotherapy. In 2013, Lima et al. used infrared thermal blankets to provide thermal vasodilation and as a result, it was found to reduce vascular resistance. Therefore, FORCLAZ brand blanket, also known as emergency blanket, used in natural disaster management, peripheral vascular resistance studies and hypothermia prevention studies was used in this study.
  Arms: Thermal Blanket Intervention Group

SUMMARY:
Peripheral arterial disease is one of the most common clinical conditions associated with cardiovascular morbidity and increased mortality, requiring exercise, antiaggregant and surgical revascularization therapy. As in peripheral arterial surgery, postoperative hypothermia is common in patients who have undergone surgical intervention and the duration of surgery is longer than 30 minutes due to the low temperature of the surgical environment or the suppression of the thermoregulation center by anesthetics and sedatives. With hypothermia, heat loss increases,peripheral vasoconstriction with activation of the sympathetic system, impaired perfusion at the surgical wound site, hypoxemia, coagulopathy, bleeding, postoperative pain, deterioration of thermal comfort, deterioration of patient comfort and prolonged hospital stay are reported. Many heating methods are used to achieve and maintain normal body temperature in the postoperative period, to prevent complications caused by hypothermia.Aluminum-coated thermal blankets are especially preferred. In this way, heat preservation, peripheral vasodilation and perfusion with the effect of temperature, reduction of muscle spasm with increased endorphin release, less pain, and increased comfort of the patient are provided. The thermal blanket is an easy-to-apply material that does not require any tools or electricity for its effectiveness and can come into direct contact with the patient's skin. It provides thermal insulation with its ability to reflect thermal radiation. Peripheral vasodilation and decreased peripheral vascular resistance have been observed with thermal therapy provided by thermal blankets. It is known that thermal blanket methods are used to warm patients in practice. However, the lack of a literature study on the regional effect of these applications on the patient has been noticed. For this purpose, in this study, the regional efficacy of thermal blankets on the patient was evaluated in order to reduce the narrowed arterial lumen and increased peripheral vascular resistance in peripheral arterial diseases and to prevent the vasoconstrictive effect of hypothermia on peripheral vessels. It was predicted that these blankets would maintain heat, increase tissue perfusion with peripheral vasodilation effect, facilitate circulation, reduce pain and facilitate mobilization.In line with this aim, the objectives are;

* To increase peripheral tissue perfusion and decrease neurovascular damage by using thermal blankets for heating after peripheral arterial surgery.
* To reduce the degree of surgical wound site and ischemic pain by using thermal blankets for warming after peripheral arterial surgery.
* To increase the patient's postoperative mobility and mobilization by using thermal blankets in peripheral artery postoperative warming.
* To contribute to the control of pain, neurovascular follow-up and reduction of damage and mobilization, which are the main nursing goals after surgery.
* To increase the comfort of the patient by utilizing the heat insulation and flexible effect of thermal blankets, thus providing an easy-to-apply, effective care in terms of nursing and increasing the quality of health care service.

Research Design This study is a randomized controlled trial to determine the effect of a thermal blanket applied to the area after peripheral arterial surgery on the patient's circulation, pain and mobilization.

DETAILED DESCRIPTION:
The population of the study consisted of patients who were planned to undergo peripheral artery surgery under elective conditions in the Cardiovascular Surgery Clinic of Seyrantepe Hamidiye Etfal Training and Research Hospital between 2022 and 2024. The sample consisted of a total of 60 patients who would undergo interventional peripheral arterial surgery, met the study criteria and agreed to participate in this study. They will be divided into two groups as 30 experimental group and 30 control group by randomization method. Data will be collected by Patient Identification Form, Visual Analog Scale (VAS-Visual Analog Scale), Neurovascular Identification Form, Patient Mobility Scale and Observer Mobility Scale.

In the implementation phase of the study, intensive care and clinical nurses will be informed about this study after obtaining institutional permission. Before the study, the patients will be informed by the researcher and after the written consent of the patients who meet the criteria for participation in the study and accept the study is obtained with the "Informed Voluntary Consent Form", respectively;

* The patient will be diagnosed with the Patient Identification Form.
* After the admission of the patient in the postoperative intensive care unit and the vital signs will be stabilized.
* General body heating of both patient groups will be done with the hot air blowing system (Forced-air), which is an active heating method.
* In the intervention group, a digital temperature probe will be fixed to the treated area just before the application of the thermal blanket (30th minute of active heating) and the temperature will be monitored for 24 hours.
* In the 30th minute of the active heating method, a thermal blanket will be applied to the treated area (extremity) of the intervention group and this application will remain for 24 hours. In the control group, cotton dressings routinely used by the clinic will be used.
* The first 24 hours after application of the thermal blanket;

  * every hour for the first 8 hours,
  * every 2 hours for the second 8 hours,
  * In the last 8 hours, pain will be evaluated every 4 hours with VAS Pain Scale and circulation will be evaluated with Neurovascular Diagnostic Form in both groups.
* At the end of the 8th hour of the thermal blanket application, the patient's first mobilization will be evaluated in both groups with the Patient Mobility and Observer Mobility Scale.
* At the end of the 24th hour of the thermal blanket application, the second mobilization assessment of the patient will be made in both groups with the Patient and Observer Mobility Scale together with pain and circulation.
* 24 hours after surgery, both groups will be transferred to the Cardiovascular Surgery Clinic without any application.
* On the second postoperative day, pain, circulation with the neurovascular diagnostic form and mobilization with the Patient and Observer Mobility Scale will be evaluated every 12 hours in both groups.
* At the end of 48 hours, mobilization will be evaluated for the last time with the Patient Mobility and Observer Mobility Scale.

The data obtained in the study will be analyzed using SPSS(Statistical Package for Social Sciences) for Windows 22.0 program.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Performing peripheral arterial surgery
* BMI<30
* No verbal communication barrier

Exclusion Criteria:

* Presence of orthopedic disability in the extremity undergoing the surgical procedure,
* Having a neurological disease
* Lack of pain control

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
The Effect of Thermal Blanket Applied to the Area After Peripheral Artery Surgery on Circulation | After applying a thermal blanket to the area, 1.2.3.4.5.6.7.8.10.12.14.16.20.24.36.48 hours
  After peripheral arterial surgery, there is a difference between the circulatory function of patients with and without thermal blankets. Circulation will be assessed 16 times with the neurovascular diagnostic form (NVT) scale in patients with thermal blankets postoperatively. Among the sub-parameters of the neurovascular diagnosis scale; skin color of the extremity (pink / red / pale / cyanotic), capillary filling time (less than 3-5 seconds), skin temperature (warm / hot / cold), pulse (strong / weak), edema (+ edema / + + + edema / absent), pain (present / absent), sensation (normal / numb / no sensation) and movement (normal / limited / no movement) will be examined. Normal findings include pink skin color and warm skin temperature, movement of extremities and fingers, tactile perception without numbness or tingling, strong and easily palpable pulses, capillary refill returning within 3-5 seconds, and absence of pain and edema.

SECONDARY OUTCOMES:
The Effect of Thermal Blanket Applied to the Area After Peripheral Artery Surgery on Pain | After applying a thermal blanket to the area, 1.2.3.4.5.6.7.8.10.12.14.16.20.24.36.48 hours
  There is a difference between the pain levels of patients with and without a thermal blanket applied to the area after peripheral arterial surgery. Pain was evaluated 16 times with the VAS (Visual Analog Scale) scale in patients who were applied a thermal blanket to the area after peripheral arterial surgery. Patients were asked to mark on a 10 cm long ruler to evaluate their pain. The distance between the point they marked and no pain is recorded in centimeters. Accordingly, "0" indicates no pain, while the average VAS value of 1-4 indicates mild pain, 5-6 indicates moderate pain, and 7-10 indicates severe pain.

OTHER OUTCOMES:
The Effect of Thermal Blanket Applied to the Area After Peripheral Artery Surgery on Mobilization | After applying a thermal blanket to the area, 8.24.48 hours
  There is a difference between the mobilization status of patients with and without thermal blanket application after peripheral arterial surgery. To evaluate this difference, the mobilization of the patient will be evaluated with the Patient Mobility and Observer Mobility Scale at the 8th hour, 24th hour and 48th hour of the thermal blanket application. For each activity, patients are asked two subgroups of questions. The answers to the questions are five-point Likert-type responses that measure the level and severity of pain perception. The increase in the scale score for the answers to the questions indicates an increase in pain and difficulty related to the activity. In the second part, 4 activities for turning, sitting, standing and walking are scored by the observer. An increase in the score indicates that the patients' mobility skills are inadequate, while a decrease in the score indicates that their mobility is good/adequate after surgical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: BIRGUL AYDOGAN, RN, Principal Investigator — Saglik Bilimleri University
Locations (1):
- Sağlık Bilimleri University, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim M, Kim EM, Oh PS, Lim ST, Sohn MH, Song EK, Park KU, Kim JY, Won KS, Jeong HJ. Usefulness of cyclic thermal therapy and red blood cell scintigraphy in patients with chemotherapy-induced peripheral neuropathy. Korean J Pain. 2021 Oct 1;34(4):427-436. doi: 10.3344/kjp.2021.34.4.427. PMID 34593660
- [Background] Simegn GD, Bayable SD, Fetene MB. Prevention and management of perioperative hypothermia in adult elective surgical patients: A systematic review. Ann Med Surg (Lond). 2021 Nov 14;72:103059. doi: 10.1016/j.amsu.2021.103059. eCollection 2021 Dec. PMID 34840773
- [Background] Torossian A, Van Gerven E, Geertsen K, Horn B, Van de Velde M, Raeder J. Active perioperative patient warming using a self-warming blanket (BARRIER EasyWarm) is superior to passive thermal insulation: a multinational, multicenter, randomized trial. J Clin Anesth. 2016 Nov;34:547-54. doi: 10.1016/j.jclinane.2016.06.030. Epub 2016 Jul 17. PMID 27687449
- [Background] Lima MV, Ochiai ME, Vieira KN, Scipioni A, Cardoso JN, Munhoz RT, Morgado PC, Barretto AC. Thermal vasodilation using a portable infrared thermal blanket in decompensated heart failure. Int Heart J. 2014;55(5):433-9. doi: 10.1536/ihj.14-096. Epub 2014 Jul 28. PMID 25070123
- [Background] Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, Collet JP, Czerny M, De Carlo M, Debus S, Espinola-Klein C, Kahan T, Kownator S, Mazzolai L, Naylor AR, Roffi M, Rother J, Sprynger M, Tendera M, Tepe G, Venermo M, Vlachopoulos C, Desormais I, Document Reviewers, Widimsky P, Kolh P, Agewall S, Bueno H, Coca A, De Borst GJ, Delgado V, Dick F, Erol C, Ferrini M, Kakkos S, Katus HA, Knuuti J, Lindholt J, Mattle H, Pieniazek P, Piepoli MF, Scheinert D, Sievert H, Simpson I, Sulzenko J, Tamargo J, Tokgozoglu L, Torbicki A, Tsakountakis N, Tunon J, Vega de Ceniga M, Windecker S, Zamorano JL. Editor's Choice - 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2018 Mar;55(3):305-368. doi: 10.1016/j.ejvs.2017.07.018. Epub 2017 Aug 26. No abstract available. PMID 28851596
- [Background] Gerhard-Herman MD, Gornik HL, Barrett C, Barshes NR, Corriere MA, Drachman DE, Fleisher LA, Fowkes FG, Hamburg NM, Kinlay S, Lookstein R, Misra S, Mureebe L, Olin JW, Patel RA, Regensteiner JG, Schanzer A, Shishehbor MH, Stewart KJ, Treat-Jacobson D, Walsh ME. 2016 AHA/ACC Guideline on the Management of Patients With Lower Extremity Peripheral Artery Disease: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2017 Mar 21;135(12):e726-e779. doi: 10.1161/CIR.0000000000000471. Epub 2016 Nov 13. PMID 27840333
- [Background] Olin JW, White CJ, Armstrong EJ, Kadian-Dodov D, Hiatt WR. Peripheral Artery Disease: Evolving Role of Exercise, Medical Therapy, and Endovascular Options. J Am Coll Cardiol. 2016 Mar 22;67(11):1338-57. doi: 10.1016/j.jacc.2015.12.049. PMID 26988957
- [Background] Seretny M, Colvin LA. Pain management in patients with vascular disease. Br J Anaesth. 2016 Sep;117 Suppl 2:ii95-ii106. doi: 10.1093/bja/aew212. PMID 27566812
- See also: Turkish Society of Cardiovascular Surgery National Society of Vascular and Endovascular Surgery Phlebology Society.(2021). National Treatment Guide for Peripheral Artery and Vein Diseases. — http://www.flebolojidernegi.org.tr/doc/ulusal_tedavi_klavuzu_2021.pdf
- See also: ESC Diagnosis of Peripheral Arterial Diseases and Treatment Guidelines — http://jag.journalagent.com/tkd/pdfs/TKDA_40_50_5_60.pdf